CLINICAL TRIAL: NCT06434740
Title: The Efficacy and Safety of Stereotactic Radiotherapy Combined With Puterizumab in Non Small Cell Lung Cancer With Intrapulmonary Metastasis：A Phase II Prospective Single Arm Clinical Study
Brief Title: A Study of SBRT Combined With Puterizumab in Intrapulmonary Metastasis From NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRS-LCsbrt
Record Dates: First submitted 2024-05-19; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: lung cancer; radiotherapy; immunotherapy; single-cell sequencing; SBRT; peripheral blood mononuclear cell; minimalResidual disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): The enrolled subjects will receive SBRT treatment combined with Puterizumab.
  Interventions: Radiation: Stereotactic Body Radiation Therapy，SBRT; Drug: Puterizumab

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy，SBRT — The enrolled subjects will receive SBRT treatment for lung metastases.The dose segmentation is 10Gy/f, with a total dose of 50Gy/5f, once every other day.
Drug: Puterizumab — Within 7-14 days after SBRT, Puterizumab should be used (dosage: recommended dosage of 200mg, intravenous infusion, infusion time of 60 minutes (± 15 minutes), once every 3 weeks (Q3W), for 6-8 months or intolerable toxicity).

SUMMARY:
This study aims to evaluate the efficacy and safety of SBRT combined with Puterizumab immunotherapy for non-small cell lung cancer with pulmonary metastases, and to determine the correlation between MRD and treatment efficacy. Through single-cell sequencing and spatial transcriptome information analysis, the underlying mechanisms will be analyzed to provide a basis for improving the new precision treatment methods for tumor immunotherapy resistance.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18
2. Non small cell lung cancer patients who have experienced pulmonary metastasis after PD-1 immunotherapy in the past
3. Voluntarily participate in this study and sign an informed consent form
4. The presence of evaluable size and number of pulmonary metastases on chest CT
5. There are indications for lung puncture biopsy
6. General physical condition (ECOG) 0-1
7. The laboratory test meets the following standards: white blood cell count>3.5 × 109/L, absolute value of neutrophils>1.8 × 109/L, platelet count ≥ 75 × 109/L, hemoglobin ≥ 100g/L; NR ≤ 1.5, and APTT ≤ 1.5 times the upper limit of normal value or partial prothrombin time (PT) ≤ 1.5 times the upper limit of normal value; Total bilirubin ≤ 1.25 times the upper limit of normal value; ALT and AST<5 times the upper limit of normal values; 24-hour creatinine clearance rate>50mL/min or blood creatinine<1.5 times the upper limit of normal value.

Exclusion Criteria:

1. Unable to tolerate or refuse further immunotherapy
2. Vulnerable groups, including individuals with mental illness, cognitive impairment, critically ill patients, minors, pregnant women, illiteracy, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
tumor response rate | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted 3 weeks and every 3 months after SBRT for up to 48 months.
  The tumor response rate will evaluate the local control of lung metastases，referring to the evaluation criteria for solid tumor efficacy RECIST 1.1

SECONDARY OUTCOMES:
Minor Residual Lesions | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted 3 weeks and every 3 months after SBRT for up to 48 months.
  Using the minimal residual disease (MRD) panel for ctDNA molecular residual detection, and through ctDNA multi-node assessment, we can dynamically monitor the therapeutic efficacy and disease recurrence.
progression-free survival | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted 3 weeks and every 3 months after SBRT for up to 48 months.
  PFS is the time from enrollment to tumor progression or death.
overall survival | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted 3 weeks and every 3 months after SBRT for up to 48 months.
  OS is the time from enrollment to death due to any reason.
RTOG acute radiation injury grading | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted during the entire SBRT process and monthly after SBRT for up to 12 months.
  Refer to the acute radiation injury grading standards of the United States Collaborative Group on Tumor Radiotherapy (RTOG)
QLQ-30 score | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted 3 weeks and every 3 months after SBRT for up to 48 months.
  The quality of life will be evaluated using the QLQ-30 score.
Lymphocyte subpopulation analysis | From the date of enrollment until the first record of tumor progression or any cause of death (whichever comes first), evaluations will be conducted 3 weeks and every 3 months after SBRT for up to 48 months.
  Using flow cytometry to detect the count and percentage of lymphocytes, including CD3+, CD3+, CD4+, CD3+, CD8+, CD4+/CD8+, and CD3-CD56+.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Sun, Ph D, Study Chair — Sir Runrun Shaw Hospital

IPD SHARING:
Plan to Share IPD: No
After the research is completed, the statistical results will be published as an article.